CLINICAL TRIAL: NCT03126851
Title: Identifying "Best Practices" for the Safe Use of Pediatric Cough and Cold Medications
Brief Title: Promoting Safe Use of Children's Cough/Cold Medicines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-01510
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Drug Labeling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No age range / no explicit warning (Experimental): Label: No age range and no explicit warning on front display panel of medication box.
  Interventions: Other: Label
- age range / no explicit warning (Experimental): Label: Age range present but no explicit warning on front display panel of medication box.
  Interventions: Other: Label
- age range / explicit warning in words (Experimental): Label: Age range present with explicit warning in words on front display panel of medication box.
  Interventions: Other: Label
- age range / explicit warning+pictogram (Experimental): Label: Age range present with explicit warning in words plus pictographic warning on front display panel of medication box.
  Interventions: Other: Label

INTERVENTIONS:
Other: Label — Labels vary based on presence or absence of age range information, and inclusion of an explicit warning in words, with or without a pictographic icon.

SUMMARY:
This study seeks to identify ways to help parents safely use cough/cold medications with their children. The study focuses on 3 key tasks that have been found to be difficult for parents: 1) decision-making about whether medicines should be given based on a child's age, 2) use of active ingredient information to determine which medications are safe to give together, and 3) medication dosing.

Specific ways that labels and dosing tools can be changed to improve parent understanding and ability to use pediatric cough and cold medications will be tested. This includes looking at whether including age restriction information on the front panel helps parents make better decisions about whether a medication should be given to a child, as well as whether presence of a specific warning or pictogram can help improve this understanding. In addition, the role of font size, including a box around ingredients, and use of a specific warning to look at and compare active ingredients, will be examined to see if these can help parents decide if two medications can be given together safely. Finally, dosing charts with pictograms of dosing tools, and provision of certain dosing tools, can lead to fewer parent dosing errors.

A label/dosing tool combination that incorporates what is learned from the first part of the study will be developed based on findings from the first part of the study, and then tested to see whether this improves parent understanding and use of pediatric cough and cold medicines.

Hypotheses include: 1) changes in labels and dosing tools, such as including explicit warnings, and pictographic warnings/instructions can improve parent understanding and ability to act on of medication instructions, 2) parents with low health literacy and/or LEP will especially benefit from strategies such as explicit wording, warnings, and pictogram, and 3) parents receiving the comprehensive labeling and dosing strategy will have a better understanding of appropriate use of cough/cold medications, including fewer dosing errors, compared to standard labels.

A multi-part experiment will be conducted. Findings will be merged with known evidence around health literacy best practices to develop a comprehensive, consumer-centered strategy for English and Spanish-speaking parents. Pilot testing of the comprehensive strategy in comparison to existing labels will then take place.

DETAILED DESCRIPTION:
See Brief summary.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Legal guardian 18 years or older
* Parent/Legal guardian with children <6 years old
* English or Spanish speaking

Exclusion Criteria:

* Visual acuity worse than 20/50 (Rosenbaum Pocket Screener)
* Uncorrectable hearing impairment
* Parents/ children too ill to participate will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
# of parents making correct decision about whether medication should be given based on age restriction information (survey) | on day of enrollment (all assessments performed on day of enrollment; study subjects will be enrolled over ~1 year period)
  # of parents making correct decision about whether medication should be given to their child based on age restriction information, assessed by survey question

SECONDARY OUTCOMES:
# of parents with correct knowledge of age group that medication can be given to (survey) | on day of enrollment (all assessments performed on day of enrollment; study subjects will be enrolled over ~1 year period)
  # of parents with correct knowledge of the age of the youngest and oldest child the medication can be given to, assessed by survey questions

CONTACTS AND LOCATIONS:
Overall Officials: Shonna Yin, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided